



## Instituto Nacional de Cardiología Ignacio Chávez

Renacimiento de la Excelencia

PROJECT TITLE: "The effect of a plant-based diet on active

rheumatoid arthritis activity"

**DOCUMENT DATE:** July 22, 2021





## Instituto Nacional de Cardiología Ignacio Chávez

Renacimiento de la Excelencia

## LETTER OF INFORMED CONSENT.

The purpose of this consent form is to provide the participants in this research with a clear explanation of its nature, as well as their role within it as participants.

This research is conducted by Dr. Fausto Sánchez Muñoz, at the Instituto Nacional de Cardiología "Ignacio Chávez". The aims of this study are to see if there is an improvement in disease activity (Rheumatoid Arthritis) with a plant-based diet.

If you agree to participate in this study, you will be asked to make a dietary change for 14 days; blood tests will be taken at the beginning and at the end of the intervention; weight and height measurements will be taken by bioimpedance; and you will receive telephone follow-up.

Participation in this study is strictly voluntary. The information collected will remain confidential and will not be used for any other purpose outside of this research. The information will be coded using an identification number and will therefore be anonymous. If you have any questions about this project, you can ask questions at any time during your participation in it. Likewise, you can withdraw from the project at any time without being harmed in any way. If at any time you notice any symptoms or complications during the dietary intervention, you should let them know.

| I voluntarily agree to participate in the study: |
|--------------------------------------------------|
| Patient name and signature: |
| Patient number: |
| Name and signature of the investigator: |
| Name and signature of witness 1: |
| Telephone and address: |
| Name and signature of witness 2: |
| Telephone and address: |